CLINICAL TRIAL: NCT06849609
Title: An Open, Dose-Escalation Early Phase Clinical Study to Evaluate the Tolerability, Safety, and Efficacy of Intrathecal of VGN-R13 in Patients with Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate the Tolerability, Safety and Efficacy of VGN-R13 in Patients with ALS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hong Chen (Other)
Responsible Party: Sponsor-Investigator, Hong Chen, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGN-R13-001
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VGN-R13 (Experimental): Up to two sequential VGN-R13 dose levels are planned. Each subject will receive one-time administration of VGN-R13 through intrathecal injection.
  Interventions: Biological: VGN-R13

INTERVENTIONS:
Biological: VGN-R13 — An adeno-associated viral vector 9 gene therapy product.

SUMMARY:
The purpose of this trial is to evaluate safety and efficacy of intrathecal delivery of VGN-R13 as a treatment of Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
The study will evaluate safety and efficacy of gene therapy in Amyotrophic Lateral Sclerosis (ALS) patients. ALS is a fatal central nervous system neurodegenerative disease. There is no effective treatment for ALS and current drug therapy has been unsuccessful in stabilizing or reversing this disease. Only supportive care is currently possible.

This study consists of screening period, treatment period and follow-up period. Eligible subjects will be enrolled. The day of administration set to be D1. Prophylactic immunosuppressive therapy will be initiated on D1. During the follow-up period (up to 52 weeks after administration), all the examinations will be completed based on the evaluation time point specified in the Schedule of Assessments table for efficacy and safety assessments until the End of Trial. Unscheduled visits may occur if the PI determines that they are necessary.

ELIGIBILITY:
key Inclusion Criteria:

1. Fully understand the purpose and risks of the study and voluntarily provide a signed and dated informed consent form.
2. Aged ≥18 years, male or female;
3. A diagnosis of ALS according to the World Federation of Neurology El Escorial criteria (revised according to the Airlie House Conference 1998 [Brooks 2000]), and confirmed through genetic diagnosis to exclude pathogenic mutations in the superoxide dismutase 1 (SOD1) and/or FUS genes;
4. The duration of the disease from the first symptom (any ALS symptom) prior to the screening must be less than 2 years (inclusive);
5. Forced Vital Capacity (FVC) adjusted for gender, age, and height (sitting position) ≥50% of the predicted value.
6. Discontinued riluzole for more than five half-lives prior to screening (and is not expected to resume during the study) or has been on a stable dose of riluzole for ≥30 days and continue to maintain this dose during the study period.
7. Discontinued edaravone for more than five half-lives prior to screening (and is not expected to resume edaravone during the study) or is receiving the standard edaravone treatment regimen at screening and has maintained a stable dose for ≥60 days (two treatment cycles) prior to administration, and continue to maintain this dose during the study period.

Key Exclusion Criteria:

1. There are other diseases related to motor neuron dysfunction (progressive bulbar palsy, primary lateral sclerosis, cervical spondylosis, lumbar spondylosis, etc., idiopathic inflammatory myopathy), which may confuse or cover up the diagnosis of ALS.
2. Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that is not managed optimally and could place a participant at an increased risk for intraoperative or postoperative bleeding. These could include, but are not limited to, anatomical factors at or near the LP site (e.g., vascular abnormalities, neoplasms, or other abnormalities) and underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., hemophilia, Von Willebrand's disease, liver disease).
3. Current severe liver or kidney or cardiovascular disease or coagulation dysfunction, autoimmune deficiency, or uncontrolled autoimmune disease or need immunosuppressive long-term treatment, poorly controlled diabetes (HBA1C ≥7% at screening) or high blood pressure, presence of sever gastrointestinal ulcers or history of gastrointestinal bleeding;
4. Presence of active infection that needs system treatment;
5. Presence or history of malignant tumors within 5 years prior to screening;
6. Significant cognitive impairment, clinical dementia, or unstable psychiatric illness, including psychosis, suicidal ideation, suicide attempt, or untreated major depression ≤ 90 days, as determined by the Investigator.
7. Current using medications including, drugs, herbal or OTC medications that strongly inhibit or induce CYP3A4 or P-glycoprotein (P-gp), e.g., metoclopramide, grapefruit juice, ketoconazole, erythromycin;
8. Received another drug for the treatment of ALS disease (including but not limited to sodium phenylbutyrate (PB), taurine diol (TURSO), tauroursodeoxycholic acid (TUDCA) within 1 month before the first dose) or ursodeoxycholic acid (UDCA), biologics or Other investigational drugs with a discontinuation period shorter than five half-lives;
9. Anticipated need, in the opinion of the Investigator, for administration of any antiplatelet or anticoagulant medication (e.g., clopidogrel) for 7 days before or 48 hours after an LP；
10. Received systemic immunosuppressive therapy within 3 months prior to screening;
11. Presence of an implanted shunt for the drainage of CSF or an implanted CNS catheter；
12. Presence of an implanted shunt for the drainage of CSF or an implanted CNS catheter；
13. Participation in gene therapy or stem cell transduction therapy at any time prior to screening；
14. Positive test result for HIV, positive treponemal antibody for syphilis, Active hepatitis B or hepatitis C infection, Active tuberculosis infection;
15. Clinically significant abnormalities in hematology or clinical chemistry parameters, as determined by the Investigator, which would render the participant unsuitable for enrollment;
16. Clinically significant, as determined by the Investigator, 12-lead ECG abnormalities, including corrected QT interval using Fridericia's correction method of > 450 ms for males and > 470 ms for females;
17. History of systemic hypersensitivity reaction to investigational product, the excipients contained in the formulation, or prophylactic immunosuppressant;
18. Contraindicated use of corticosteroids and sirolimus;
19. History of drug abuse or alcoholism within ≤ 6 months of study enrollment that would limit participation in the study, as determined by the Investigator;
20. Alcohol abuse (drinking more than 14 units of alcohol per week) or smoking more than 5 cigarettes per day on average in the 6 months prior to screening;
21. Pregnant or breastfeeding women;
22. Other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the participant unsuitable for enrollment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | up to 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.

SECONDARY OUTCOMES:
Change From Baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Total Score | up to 52 weeks
  The ALSFRS-R measures 4 functional domains, including respiratory, bulbar function, gross motor skills, and fine motor skills. There are 12 questions, each scored from 0 (no function) to 4 (full function), for a total possible score of 48. Scores decline with disease progression. ALSFRS-R scores calculated at diagnosis can be compared to scores throughout time to determine the speed of progression. Higher scores represent better function, negative change from baseline indicates disease progression.
Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) | up to 52 weeks
  Vital capacity is measured by means of an FVC test.
Time to Death or Permanent Ventilation | up to 52 weeks
  Time to Death or Permanent Ventilation is defined as the time to the earliest occurrence of one of the following events that were adjudicated by an independent committee: Death; Permanent ventilation (≥22 hours of mechanical ventilation [invasive or noninvasive] per day for ≥21 consecutive days).
Change From Baseline in Handheld Dynamometry (HHD) Megascore as Measured by the HHD Device | up to 52 weeks
  Quantitative muscle strength is evaluated using HHD, which tests isometric strength of multiple muscles using standard participant positioning.
The antibody titer | up to 52 weeks
  Immunogenicity
Immunogenicity | up to 52 weeks
  the number of subjects with positive anti-AAV9 in the blood and CSF.

CONTACTS AND LOCATIONS:
Locations (1):
- TongJi Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGN-R13 is fully approved.